CLINICAL TRIAL: NCT04369508
Title: PD-L1-expressing Regulatory T Cells in Blood and Urine of Localized Prostate Cancer Patients Undergoing Iodine-125 Permanent Brachytherapy
Brief Title: PD-L1-expressing Regulatory T Cells in Localized Prostate Cancer Patients Undergoing Iodine-125 Permanent Brachytherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, ou tongwen, chairman of urology, Xuanwu Hospital, Beijing
Other Study IDs: 20200428003
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: permanent brachytherapy — Briefly, the patient had a general anesthesia and PPB was performed by using the "real-time" intraoperative planning method guided by TRUS. The radioactive seeds were inserted transperineally according to a modified peripherally loaded Seattle technique 17. I-125 was used for all implants with a mean seed activity of 0.45 mCi per seed. All procedures were completed by a single surgeon.

SUMMARY:
Immunotherapy is currently revolutionizing the field in oncology. However, prostate cancer is poorly responsive to immune checkpoint inhibition. The combination of immunotherapy and radiotherapy is an emerging clinical treatment aradigm. X-ray radiation treatment can activate both the adaptive and innate immune systems through directly killing tumor cells, causing mutations in tumor-derived peptides, and causing localized inflammation that increases immune cell trafficking to tumors. Recently, preclinical study reported that immune checkpoint inhibition combined with radiotherapy treats CPRC with significant increases in median survival compared to drug alone.

DETAILED DESCRIPTION:
Permanent brachytherapy is one of those standard treatments for localized prostate cancer patients.

Biopsy confirms prostate cancer. Blood and urine of localized prostate cancer patients will be collected before and at different time points after permanent brachytherapy (1, 3, 6, and 12 months)

ELIGIBILITY:
Inclusion Criteria:

- Biopsy confirms prostate cancer

Localized Prostate Cancer, ≤cT3

No chemotherapy or Hormonal therapy before Permanent Brachytherapy

Exclusion Criteria:

- Unacceptable operative risk

Poor anatomy which in the opinion of the radiation oncologist could lead to a suboptimal implant (e.g.,large or poorly healed transurethral resection of the prostate (TURP) defect, large median lobe, large gland size).

Pathologically positive lymph nodes

Significant obstructive uropathy

Distant metastases

Use steroids regularly

The diagnosis was accompanied by immune-related diseases

Allergic constitution

Abnormal white blood cell and lymphocyte counts

Ever underwent other treatments for prostate cancer, such as chemotherapy or Hormonal therapy

Accompanied by other malignancies

Splenectomy

HIV positive

Receive an anti-infective vaccine for the last 6 months

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: localized prostate cancer patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the level of PD-L1-expressing regulatory T cells in blood and urine | 2 year
  the level of PD-L1-expressing regulatory T cells in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Tongwen Ou, MD., Study Chair — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No